CLINICAL TRIAL: NCT02260869
Title: A Prospective Double Blind, Randomized Control Trial to Compare the Efficacy of Cool Radiofrequency Ablation vs. Conventional Monopolar Radiofrequency Ablation of the Geniculate Nerves for the Treatment of Chronic Osteoarthritic Knee Pain
Brief Title: Efficacy of Cooled and Monopolar Radiofrequency Ablation of the Geniculate Nerves for the Treatment of Chronic Osteoarthritic Knee Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to financial constraints, sponsor could not complete the study.
Sponsor: Millennium Pain Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MPC-2014-GNK
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Results first posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cooled radiofrequency ablation (Active Comparator): Patient is placed in supine position on a fluoroscopic table with a pillow under the popliteal fossa. An anterio-posterior fluoroscopic view of the tibio-femoral joint is obtained. Skin and subcutaneous tissues are anesthetized and a 17 g introducer needle is advanced percutaneously towards the junction of shaft with epicondyle until bone contact is made. The needle is then laterally displaced away from the bone. This process is performed at the superior medial and superior lateral aspects of the femur, and the inferior medial aspect of the tibia. The fluoroscope is placed in lateral view to guide the needle depth to be at the medial third of the femur or tibia. A cooled radiofrequency probe from a Pain Management Radiofrequency kit is advanced through the introducer. Following sensory and motor stimulation, cooled genicular nerve radiofrequency ablation is carried out at 60 Celsius for 150 seconds.
  Interventions: Procedure: Genicular nerve radiofrequency ablation; Device: Pain Management Radiofrequency Kit
- Monopolar radiofrequency ablation (Active Comparator): Patient is placed in supine position on a fluoroscopic table with a pillow under the popliteal fossa. An anterio-posterior fluoroscopic view of the tibio-femoral joint is obtained. Skin and subcutaneous tissues are anesthetized and a 16 g introducer needle is advanced percutaneously towards the junction of shaft with epicondyle until bone contact is made. The needle is then laterally displaced away from the bone. This process is performed at the superior medial and superior lateral aspects of the femur, and the inferior medial aspect of the tibia. The fluoroscope is placed in lateral view to guide the needle depth to be at the medial third of the femur or tibia. A conventional radiofrequency probe from a Pain Management Radiofrequency kit is advanced through the introducer. Following sensory and motor stimulation, genicular nerve radiofrequency ablation will be carried out at 80 Celsius for 90 seconds.
  Interventions: Procedure: Genicular nerve radiofrequency ablation; Device: Pain Management Radiofrequency Kit

INTERVENTIONS:
Procedure: Genicular nerve radiofrequency ablation — Radiofrequency ablation uses the electrical field generated by a radiofrequency probe inserted near a nerve responsible for pain. Chronic pain sensation in the knee is generated at the genicular nerves. The physician locates the affected genicular nerve by injecting an anesthetic (lidocaine) that produces a sensory nerve block (i.e. anesthetic pain relief). A radiofrequency probe is inserted percutaneously near the affected nerve using a cannula/introducer and is then connected to a radiofrequency generator. This is set to stimulate sensory and motor response, which allows the physician to adjust the probe position for effective and safe treatment. Then radiofrequency is applied to the tissue for a short time (up to 150 seconds) in order to generate a target temperature (no more than 80 degrees Celsius). The increase in the temperature of the tissue ablates the affected nerve producing pain relief.
  Other Names: genicular neurotomy using radiofrequency
Device: Pain Management Radiofrequency Kit — The pain management radiofrequency consists of a radiofrequency generator, a radiofrequency probe and an introducer/cannula. The introducer cannula is used to percutaneously position the probe in the appropriate location for treatment. The radiofrequency probe is an electrode that delivers the electric field that heats up the tissue. In cooled radiofrequency the electrode is surrounded by a water jacket that cools it while heat is generated. The generator is the instrument that provides the radiofrequency according to a particular temperature and time program. Temperature, tissue impedance and radiofrequency power are lalso monitored by the generator.

SUMMARY:
This is a single center randomized controlled trial. Approximately 102 patients will be randomized to one of two treatment groups: cooled radiofrequency or conventional monopolar radiofrequency ablation. Patients with chronic knee pain, with moderate to severe osteoarthritis according to the Kellgren-Lawrence scale for at least 6 months who have failed conservative therapy will be screened for the study.

Then, patients will be enrolled based on reporting ≥50% pain relief after a fluoroscopic guided single diagnostic block of the geniculate nerves (superior medial, superior lateral, and inferior medial) with 0.5 ml of local anesthetic (2% Lidocaine).

Baseline data will be collected for all enrolled patients. Outcomes will be measured at 1, 4, 12, 24 and 52 weeks.

Outcome measures will be: Visual analogue scale (VAS) both while at rest and during ambulation, Oxford knee scores, WOMAC, and global perceived effect.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have given their written informed consent to participate in this clinical study based on voluntary agreement after a thorough explanation of the patient's participation is provided to them.
* Female patients who are not pregnant and do not plan to become pregnant during the study. Females of child bearing potential must provide a negative pregnancy test provided by the study physician and must be using reliable contraception and must continue to use reliable contraception until study completion at 52 weeks. Non-childbearing potential is defined as postmenopausal for at least 2 years or surgical sterilization or hysterectomy at least 3 months before study start.
* Must be older than 18 years old..
* Must have chronic knee pain for at least 6 months.
* Must have radiologic evidence of OA of the knee, grade 2-4 based on the Kellgreen-Lawrence scale.
* Persistent pain despite the use of conservative treatment (physical therapy, oral analgesic, steroid injections).
* Must have a VAS score of at least 5 with ambulation.
* Subjects must be on a stable dose of pain medication regimen for at least 2 months.
* Greater than or equal to 50% improvement from blocks in target knee for duration of the anesthetic.

Exclusion Criteria:

* Knee pain must not be acute.
* Previous total knee replacement.
* Evidence of connective tissue disease.
* Patients who have a BMI greater than 40.
* Evidence of serious neurological or psychiatric disorders.
* Current opioid use must not be greater than or equal to 90 mg morphine equivalent per 24 hour period.
* Must not have radicular pain in the affected limb.
* Patients with uncorrected coagulation disorders or who are on anticoagulation therapy and cannot interrupt the therapy.
* Patients who have pacemakers or generators.
* Patient who are pregnant, breast-feeding or women of childbearing potential with positive pregnancy tests.
* Sexually active female patients of childbearing potential who are not willing to use adequate contraceptive measures to avoid pregnancy until week 52 of the study. Sexually active male patients who are not willing to use adequate contraceptive measures until week 52 of the study. Adequate methods of birth control include the following: Hormonal contraception (female patients) or use of at least one acceptable double-barrier method (for example: diaphragm plus spermicidal agent or condoms (male or female) plus spermicidal agent.), vasectomy, intrauterine device, and/or exclusive sexual partner for whom one of the above acceptable methods applies.
* Patients who have cancer or a past history of any cancer within 5 years prior to the time of informed consent, with the exception of basal cell or squamous cell carcinoma of the skin.
* Human immunodeficiency virus (HIV) infection or a clinically significant infection.
* A clinically significant disorder such as cerebrovascular disease, pulmonary infarction, ischemic heart disease, cardiac dysrhythmia, myocardial infarction, or congestive heart failure.
* Uncontrolled diabetes, uncontrolled pulmonary disease, or uncontrolled hypertension.
* Patients who have evidence of major psychiatric disease, mental disorder, drug dependency, alcohol dependency, or substance abuse disorders.
* Any patient with a medical condition and/or disease that the Investigator believes could affect the study results or the safe conduct of the study.
* Patients who are receiving compensation according to Workers' Compensation Act or are involved in personal injury litigation.
* Patients who participated in another clinical study within 3 months prior to the time of informed consent, or who are expected to participate in another study during the period of this study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2019-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Vallejo, MD, PhD, Principal Investigator — Millennium Pain Center
Locations (3):
- United States (3):
  - Millennium Pain Center, Bloomington, Illinois
  - Millennium Pain Center at Decatur Memorial Hospital, Decatur, Illinois
  - Methodist Comprehensive Spine and Pain Center - Millennium Pain Center, Peoria, Illinois

REFERENCES:
- [Background] Murphy L, Helmick CG. The impact of osteoarthritis in the United States: a population-health perspective: A population-based review of the fourth most common cause of hospitalization in U.S. adults. Orthop Nurs. 2012 Mar-Apr;31(2):85-91. doi: 10.1097/NOR.0b013e31824fcd42. PMID 22446800
- [Background] Jordan JM, Helmick CG, Renner JB, Luta G, Dragomir AD, Woodard J, Fang F, Schwartz TA, Abbate LM, Callahan LF, Kalsbeek WD, Hochberg MC. Prevalence of knee symptoms and radiographic and symptomatic knee osteoarthritis in African Americans and Caucasians: the Johnston County Osteoarthritis Project. J Rheumatol. 2007 Jan;34(1):172-80. PMID 17216685
- [Background] Peat G, McCarney R, Croft P. Knee pain and osteoarthritis in older adults: a review of community burden and current use of primary health care. Ann Rheum Dis. 2001 Feb;60(2):91-7. doi: 10.1136/ard.60.2.91. PMID 11156538
- [Background] Karaman H, Tufek A, Kavak GO, Yildirim ZB, Uysal E, Celik F, Kaya S. Intra-articularly applied pulsed radiofrequency can reduce chronic knee pain in patients with osteoarthritis. J Chin Med Assoc. 2011 Aug;74(8):336-40. doi: 10.1016/j.jcma.2011.06.004. Epub 2011 Jul 23. PMID 21872812
- [Background] Choi WJ, Hwang SJ, Song JG, Leem JG, Kang YU, Park PH, Shin JW. Radiofrequency treatment relieves chronic knee osteoarthritis pain: a double-blind randomized controlled trial. Pain. 2011 Mar;152(3):481-487. doi: 10.1016/j.pain.2010.09.029. Epub 2010 Nov 4. PMID 21055873
- [Background] Ikeuchi M, Ushida T, Izumi M, Tani T. Percutaneous radiofrequency treatment for refractory anteromedial pain of osteoarthritic knees. Pain Med. 2011 Apr;12(4):546-51. doi: 10.1111/j.1526-4637.2011.01086.x. Epub 2011 Apr 4. PMID 21463469
- [Background] Vallejo R, Benyamin R, Tilley DM, Kelley CA, Cedeno DL. An ex vivo comparison of cooled-radiofrequency and bipolar-radiofrequency lesion size and the effect of injected fluids. Reg Anesth Pain Med. 2014 Jul-Aug;39(4):312-21. doi: 10.1097/AAP.0000000000000090. PMID 24781285

RESULTS

PARTICIPANT FLOW:
Groups:
- Cooled Radiofrequency Ablation: Radiofrequency ablation of the genicular nerves of osteoarthritic knee(s) using a cooled radiofrequency ablation probe
- Monopolar Radiofrequency Ablation: Radiofrequency ablation of the genicular nerves of osteoarthritic knee(s) using a monopolar radiofrequency ablation probe (16-gauge)
Period: Overall Study
Arm/Group | Cooled Radiofrequency Ablation | Monopolar Radiofrequency Ablation
Started | 38 | 37
Completed | 31 | 29
Not Completed | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cooled Radiofrequency Ablation | Monopolar Radiofrequency Ablation | Total
Number analyzed (Participants) | 38 | 37 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (10.3) | 56.8 (12.3) | 60.0 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 25 | 52
  Male | 11 | 12 | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 33.0 (5.2) | 31.9 (4.6) | 32.5 (5.0)
Knee Pain VAS Score [Mean (Standard Deviation); unit: mm] — The 100 mm Visual Analog Scale (VAS) was used to assess pain level by subjects. The scale consists of a 100 mm long line without marks between the 0 and 100 mm edges. Range of scale is 0 to 100 mm, where 0 means no pain and 100 mm means the worst pain imaginable.
  mm | 74.4 (12.2) | 73.0 (11.3) | 73.7 (11.7)
Oxford Knee Score [Mean (Standard Deviation); unit: oxford knee score] — The Oxford Knee Score (OKS) measures the level of function, activities of daily living and how they have been affected by knee pain over the preceding four weeks. The OKS is a obtained from a 12-item patient reported questionnaire. Each item has 5 categories, scored from 0 to 4, with 0 being the worst outcome and 4 the best outcome of each item. The OKS is the sum of all item scores. Therefore, it ranges from 0 to 48, with 0 being the worst functional outcome possible and 48 is the best functional outcome possible.
  oxford knee score | 19.9 (7.4) | 17.7 (5.2) | 18.8 (6.5)

OUTCOME MEASURES:

1. Primary Outcome: Evidence of Change in Knee Pain
Description: A 100mm visual analog scale (VAS) score at 24 weeks post-treatment will be compared to baseline score to measure change in pain level.
  Change in Pain = (VAS at 24 weeks) - (VAS at baseline) The VAS consists of a 100 mm long line without marks between the 0 and 100 mm edges. Range of scale is 0 to 100 mm, where 0 means no pain and 100 mm means the worst pain imaginable.
  A negative change in VAS means a reduction in pain level after 24-weeks of treatment.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: knees
Arm/Group | Cooled Radiofrequency Ablation | Monopolar Radiofrequency Ablation
Number analyzed (Participants) | 38 | 37
Number analyzed (knees) | 49 | 47
mm | -40.7 (26.8) | -38.6 (27.8)

2. Secondary Outcome: Evidence of Functional Changes
Description: Standard score system (Oxford Knee Score) was used to assess functional changes at 24 weeks of treatment relative to baseline. The Oxford Knee Score (OKS) measures the level of function, activities of daily living and how they have been affected by knee pain. The OKS is a obtained from a 12-item patient reported questionnaire. Each item has 5 categories, scored from 0 to 4, with 0 being the worst outcome and 4 the best outcome of each item. The OKS is the sum of all item scores. Therefore, it ranges from 0 to 48, with 0 being the worst functional outcome possible and 48 is the best functional outcome possible.
  Change in OKS = (OKS at 24 weeks) - (OKS at baseline) A positive Change in OKS indicates an improvement in extent of function.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: Oxford Knee Score
Units Other Than Participants: knees
Arm/Group | Cooled Radiofrequency Ablation | Monopolar Radiofrequency Ablation
Number analyzed (Participants) | 38 | 37
Number analyzed (knees) | 49 | 47
Oxford Knee Score | 10.7 (9.1) | 12.7 (10.4)

ADVERSE EVENTS:
Time Frame: Adverse events were collected since the start of enrollment and randomization until the 52 weeks follow up visit.
Arm/Group | Cooled Radiofrequency Ablation | Monopolar Radiofrequency Ablation
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/37
Serious Adverse Events (participants affected / at risk) | 2/38 | 4/37
Other Adverse Events (participants affected / at risk) | 18/38 | 20/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cooled Radiofrequency Ablation (N=38) | Monopolar Radiofrequency Ablation (N=37)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Broken Left Femur (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Worsening of reflux esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cooled Radiofrequency Ablation (N=38) | Monopolar Radiofrequency Ablation (N=37)
Knee Pain or Swelling (Musculoskeletal and connective tissue disorders) | 6 (8) | 4 (4)
Other pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Bruised body parts (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Respiratory tract infections (Infections and infestations) | 7 (10) | 9 (12)
Muscular issues (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3)

LIMITATIONS AND CAVEATS:
Early termination led to a number of subjects analyzed below the required statistical power to measure a significant difference between the means

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-24): https://cdn.clinicaltrials.gov/large-docs/69/NCT02260869/Prot_SAP_000.pdf